CLINICAL TRIAL: NCT05150691
Title: A Phase 1/2a, Multicenter, Open-Label, First in Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of DB-1303/BNT323 in Patients With Advanced/Metastatic Solid Tumors
Brief Title: A Phase 1/2a Study of DB-1303/BNT323 in Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DB-1303-O-1001
Record Dates: First submitted 2021-11-11; First posted 2021-12-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HER2-positive Advanced Solid Tumor
Keywords: HER2; HER2-positive; HER2-positive Breast Cancer; HER2-positive Gastric Cancer; HER2-positive Endometrial Cancer; HER2-positive Biliary Tract Cancer; HER2-positive Advanced Solid Tumor; HER2 low; HER2 high; metastatic cancer; HER2-positive GEJ; Uterine serous papillary carcinoma; USPC; recurrent cancer; carcinoma; neoplasms; breast neoplasms; gastrointestinal neoplasms; endometrial neoplasms; biliary tract neoplasms; Antineoplastic Agents, Biological; stomach cancer; bile duct cancer; Cholangiocarcinoma; liver cancer; liver neoplasms; NSCLC; Non-Small Cell Lung Cancer; NSCLC HER2 mutation; HER2 Low Breast Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Carcinoma; Neoplasms; Breast Neoplasms; Gastrointestinal Neoplasms; Endometrial Neoplasms; Biliary Tract Neoplasms; Stomach Neoplasms; Bile Duct Neoplasms; Cholangiocarcinoma; Liver Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pertuzumab; Ritonavir; Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (24):
- DB-1303/BNT323 Dose Level 1 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 at Dose Level 1 on Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Level 2 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 at Dose Level 2 on Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Level 3 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 at Dose Level 3 on Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Level 4 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 at Dose Level 4 on Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Level 5 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 at Dose Level 5 on Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 1 (Experimental): Enrolled Subjects will be randomized to receive a single-dose of DB-1303/BNT323 on a selected dose level 1 or dose level 2 Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 2 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 3 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 4 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 5 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Level 6 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 at Dose Level 6 on Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Level 7 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 at Dose Level 7 on Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 6 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 7 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 8 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 9 (Experimental): Enrolled Subjects will be randomized to receive a single-dose of DB-1303/BNT323 on a selected dose level 1 or dose level 2 on Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 10 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W along with ritonavir or itraconazole to assess the DDI potential
  Interventions: Biological: DB-1303/BNT323; Drug: Ritonavir; Drug: Itraconazole
- DB-1303/BNT323 Dose Expansion 11 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 12 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level 1 or dose level 2 in combination with Pertuzumab on Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323; Drug: Pertuzumab Injection
- DB-1303/BNT323 Dose Expansion 13 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 14 (Experimental): China Only:Subjects who were previously treated with trastuzumab and taxane will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 15 (Experimental): China Only: Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 16 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323
- DB-1303/BNT323 Dose Expansion 17 (Experimental): Enrolled Subjects will receive a single-dose of DB-1303/BNT323 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Biological: DB-1303/BNT323

INTERVENTIONS:
Biological: DB-1303/BNT323 — Administered IV
Drug: Pertuzumab Injection — Administered IV
  Arms: DB-1303/BNT323 Dose Expansion 12
Drug: Ritonavir — Administered oral
  Arms: DB-1303/BNT323 Dose Expansion 10
Drug: Itraconazole — Administered oral
  Arms: DB-1303/BNT323 Dose Expansion 10

SUMMARY:
This is a dose-escalation and dose-expansion Phase 1/2a trial to evaluate the safety and tolerability of DB-1303/BNT323 in subjects with advanced solid tumors that express HER2.

DETAILED DESCRIPTION:
This is a multicenter, non-randomized (Except for Dose Expansion 1 and Dose Expansion 9 cohorts), open-label, multiple-dose, FIH study. The study consists of two parts: Part 1 adopts an accelerated titration at first dose level followed with classic "3+3" design to identify the MTD/RP2D; Part 2 is a dose expansion phase to confirm the safety, tolerability and explore efficacy in selected malignant solid tumors at the MTD/the RP2D. This study will enroll subjects with advanced/unresectable, recurrent, or metastatic HER2-expressing malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Has a pathologically documented HER2-positive or HER2-expressing (except for cohort 2h where the requirement is HER2-null), advanced/unresectable, recurrent, or metastatic malignant solid tumor that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.
* At least 1 measurable lesion (per RECIST 1.1)
* Provide signed informed consent
* ECOG performance status (PS) of 0-1.
* LVEF ≥ 50% by ECHO or MUGA
* Adequate organ functions
* Provide pre-existing diagnosis of HER2 status or resected tumor samples or undergo fresh tumor biopsy for HER2 testing.
* Life expectancy of ≥ 3 months.

Additional Inclusion Criteria for Part 2 Expansion Group 9:

1. Has pathologically documented advanced/unresectable, recurrent, or metastatic EC (including UCS and USPC) and has progressed on or after at least 1 line of systemic treatment including platinum-based therapy and exposure to ICI but no more than prior 3 lines of therapy for advanced/unresectable, or metastatic disease. Note: endocrine therapy will not qualify as a systemic therapy line.

Exclusion Criteria:

* History of symptomatic CHF (New York Heart Association [NYHA] classes II-IV) or serious cardiac arrhythmia requiring treatment.
* History of myocardial infarction or unstable angina within 6 months before Day 1.
* Average QTcF > 450 ms in males and > 470 ms in females
* History of clinically significant lung diseases
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
* HIV infection with AIDS defining illness or active viral hepatitis.
* Clinically active brain metastases
* Unresolved toxicities from previous anticancer therapy, defined as toxicities not yet resolved to NCI-CTCAE version 5.0, Grade ≤ 1 or baseline.
* A known hypersensitivity to either the drug substances or inactive ingredients in the drug product.
* Part 2 (expansion) Only:Multiple primary malignancies within 3 years, except adequately resected non- melanoma skin cancer, curatively treated in-situ disease, other solid tumors curatively treated, or contralateral breast cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 796 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Percentage of Participants with Dose-Limiting Toxicities (DLTs) as assessed by CTCAE v5.0. | up to 21 days after C1D1
  Percentage of participants in Part 1 with DLTs
Phase 1: Percentage of participants with AEs in Part 1 graded according to NCI CTCAE v5.0 | Up to Safety Follow-Up visit, approximately 35 days post-treatment
  Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) or Treatment Emergent Adverse Event of Special Interest include those >/= G3 leading to dose reduction, interruption or discontinuation as assessed by CTCAE v5.0, abnormal vital signs, abnormal 12-lead ECGs, abnormal safety laboratory tests, abnormal ECOG PS, abnormal ECHO/MUGA (LVEF).
Phase 1: Percentage of Participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of Participants with SAEs in Part 1 graded according to NCI CTCAE v5.0
Phase 1: Maximum Tolerated Dose (MTD) of DB-1303 | Up to Safety Follow-Up visit, approximately 35 days post-treatment
  MTD on the data collected during Part 1
Phase 1: Recommended Phase 2 Dose (RP2D) of DB-1303 | Up to Safety Follow-Up visit, approximately 35 days post-treatment
  RP2D of DB-1303 based on the data collected during Part 1
Percentage of participants with AEs in Part 2 graded according to NCI CTCAE v5.0 | Up to follow-up period, approximately 1 year post-treatment
  Phase 2: Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) or Treatment Emergent Adverse Event of Special Interest include those >/= G3 leading to dose reduction, interruption or discontinuation as assessed by CTCAE v5.0, abnormal vital signs, abnormal 12-lead ECGs, abnormal safety laboratory tests, abnormal ECOG PS, abnormal ECHO/MUGA (LVEF).
Phase 2: Percentage participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with SAEs in Part 2 graded according to NCI CTCAE v5.0
Phase 2: Percentage of Objective Response Rate (ORR) as assessed by RECIST 1.1. | Up to follow-up period, approximately 1 year post-treatment
  The percentage of subjects who had a best response of CR or PR, for Part 2 only which was maintained ≥4 weeks.
Phase 2 (Dose Expansion 10 only): To evaluate the effect of ritonavir on DB-1303 and P1003 PK in subjects with HER2-expressing, HER2-amplified, or HER2-mutated advanced solid malignant tumors | up to safety follow-up visit, approx. 35 days post-treatment
  Maximum observed plasms concentration (Cmax) and Area under the concentration-time curve from 0 to infinity of DB-1303 and P1003 (+/- Ritonavir)
Phase 2 (Dose Expansion 10 only): To evaluate the effect of itraconazole on DB-1303 and P1003 PK in subjects with HER2-expressing, HER2-amplified, or HER2-mutated advanced solid malignant tumors. | up to safety follow-up visit, approx. 35 days post-treatment
  Maximum observed plasms concentration (Cmax) and Area under the concentration-time curve from 0 to infinity of DB-1303 and P1003 (+/- Itraconazole)

SECONDARY OUTCOMES:
Phase 1 & Phase 2: Pharmacokinetic-AUC | Up to safety follow up visit, approx. 35 days post-treatment
  Area under the concentration-time curve from time 0 to infinity of DB-1303
Phase 1 & Phase 2: Pharmacokinetic-Cmax | Up to safety follow up visit, approx. 35 days post-treatment
  Maximum observed plasma concentration (Cmax) of DB-1303
Phase 1 & Phase 2: Pharmacokinetic-Tmax | Up to safety follow up visit, approx. 35 days post-treatment
  Time to Cmax of DB-1303
Phase 1 & Phase 2: Pharmacokinetic-T1/2 | Up to safety follow up visit, approx. 35 days post-treatment
  Terminal elimination half-life
Phase 1 & Phase 2: Pharmacokinetic-Ctrough | Up to safety follow up visit, approx. 35 days post-treatment
  Trough concentration of DB-1303
Phase 1 & Phase 2: Pharmacodynamics-ADA | Up to safety follow up visit, approx. 35 days post-treatment
  Data gathered from blood to determine Levels of anti-drug antibody (ADA) against DB 1303 in serum compared to baseline.
Phase 1 & 2: Disease Control Rate (DCR) as assessed by RECIST 1.1 | Up to follow-up period, approximately 1 year post-treatment
  Proportion of participants who had a best response rating of CR or PR, or SD using RECIST V1.1.
Phase 1 & 2: Duration of Response (DoR) as assessed by RECIST 1.1 | Up to follow-up period, approximately 1 year post-treatment
  The duration of time from date of first CR or PR to date of progressive disease or death due to any cause, whichever comes first using RECIST V1.1
Phase 1 & 2: Time to Response (TTR) as assessed by RECIST 1.1 | Up to follow-up period, approximately 1 year post-treatment
  The duration of time when receiving the first dose of study drug to the first date that is evaluated as either CR or PR using RECIST V1.1
Phase 2: Time on Therapy | Up to 21 days after the participant's last dose
  The duration of time from participant receiving first dose of study drug to the last dose + 21 days
Phase 2: Percent change in target lesions as assessed by RECIST 1.1 | Up to follow-up period, approximately 1 year post-treatment
  The percent change in the participant's target lesions from baseline to last study scan using RECIST V1.1
Phase 1 and 2 Cohort b only: Progression-Free Survival | Up to follow-up period, approximately 1 year post-treatment
  Time from subject receiving the first dose to disease progression or death by any cause
Phase 1 and 2 Cohort b only: Overall Survival | Up to follow-up period, approximately 1 year post-treatment
  Time from subject receiving the first dose to death by any cause
Phase I: Percentage of Objective Response Rate (ORR) as assessed by investigator based on RECIST 1.1 | Up to follow-up period, approximately 1 year post-treatment
  The percentage of subjects who had a best response of CR or PR
Phase 2 Cohort b Only: Percentage of ORR as assessed by IRC and as assessed by investigator based on RECIST 1.1 for HER2-expressing subjects and in subjects with prior ICI treatment | Up to follow-up period, approximately 1 year post-treatment
  The percentage of subjects who had a best response of CR or PR, for Cohort 2b only
To evaluate the safety of DB-1303 with/without ritonavir or itraconazole | Up to follow-up period, approximately 1 year post-treatment
  Percentage of Participants with Serious Adverse Events (SAEs), Treatment Emergent Adverse Events (TEAE), TEAEs >/= G3, or TEAEs leading to dose reduction, interruption or discontinuation, Adverse Events of Special Interest, (AESIs), abnormal vital signs, abnormal 12-lead ECGs, abnormal safety laboratory tests, abnormal ECOG PS, abnormal ECHO/MUGA (LVEF).

CONTACTS AND LOCATIONS:
Locations (102):
- United States (35):
  - Helios Clinical Research, Cerritos, California
  - California Research Institute, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Advanced Research LLC, Coral Springs, Florida
  - The Oncology Institute of Hope and Innovation, Lakeland, Florida
  - D&H Cancer Research Center LLC, Margate, Florida
  - HCA Mercy Hospital, Miami, Florida
  - BRCR Medical Center Inc., Plantation, Florida
  - BRCR Medical Center Inc., Tamarac, Florida
  - Southeastern Regional Medical Center, LLC, Newnan, Georgia
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - University of Chicago, Chicago, Illinois
  - Women's Cancer Care, Covington, Louisiana
  - Holy Cross Hospital, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Profound Research LLC/Michigan Hematology & Oncology Consultants, Dearborn, Michigan
  - David C. Pratt Cancer Center, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Northwell Health, Lake Success, New York
  - Laura & Isaac Perlmutter Cancer Center at NYC Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - North Shore Hematology Oncology Associate P.C. DBA New York Cancer and Blood Specialists, Shirley, New York
  - Regional Medical Oncology Center, Wilson, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Rittenhouse Hematology Oncology, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - AHN West Penn Hospital, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Clinical Trial Network, Houston, Texas
  - Oncology and Hematology of South Texas, PA, Laredo, Texas
  - NEXT Virginia, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
- Australia (4):
  - Scientia Clinical Research LTD, Randwick, New South Wales
  - Macquarie Clinical Trials Unit, Sydney, New South Wales
  - Integrated Clinical Oncology Network Pty Ltd (Icon), South Brisbane, Queensland
  - Monash Health, Melbourne, Victoria
- China (50):
  - The first affiliated hospital of Bengbu medical college, Bengbu, Anhui
  - Anhui provincial hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - The First Hospital of Jilin University, Hongcun, Changchun
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First affiliated hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Maternity and Child-care Hospital, Lanzhou, Gansu
  - Huizhou First Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Zhongshan University, Guangzhou, Guangdong
  - The First affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First people's hospital of Yulin, Yulin, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Henan cancer Hospital, Zhengzhou, Hehan
  - Anyang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union hospital Tongji Medical college Huazhong university of science and technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Hunan People's Provincial Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Changzhou Tumor Hospital, Changzhou, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Xuzhou Cancer Hospital, Xuzhou, Jiangsu
  - Jiangxi maternal and child health hospital, Nanchang, Jiangxi
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning cancer hospital & Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Central hospital affiliated to Shandong first medical university, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer hospital & institute, Jinan, Shandong
  - Affiliated hospital of Jining medical university, Jining, Shandong
  - Linyi Tumor Hospital, Liaocheng, Shandong
  - Zibo Central hospital, Zibo, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shangdong
  - Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Tenth people's Hospital, Shanghai, Shanghai Municipality
  - The Obstetrics & Gynecology Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical university cancer institute & hospital, Tianjin, Tianjin Municipality
  - Yunnan Provincial Cancer Hospital, Kunming, Yunnan
  - 1st affliated hospital of Zhejiang University, Hangzhou, Zhejiang
  - The second affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Women's hospital school of medicine Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- BRCR Global Puerto Rico LLC., Mayagüez, Puerto Rico
- South Korea (5):
  - Seoul National University Bundang Hospital, Gyeonggi-do, Bundang-gu
  - Samsung Medical Center, Seoul, Gangnam-gu
  - National Cancer Center, Gyeonggi-do, Ilsandong-gu
  - Severance Hospital, Seoul, Seodaemun-gu
  - Asan Medical Center, Seoul, Songpa-gu
- Taiwan (7):
  - Taipei Veterans General Hospital, Taipei, Beitou District
  - Changhua Christian Hospital, Changhua, Changhua County
  - Taipei Medical University Hospital, Taipei, Xinyi District
  - Taipei Medical University-Shuang Ho Hospital, Taipei, Zhonghe District
  - Mackay Memorial Hospital-Taipei, Taipei, Zhongshan District
  - National Taiwan University Hospital, Taipei, Zhongzheng District
  - Kaohsiung Veterans General Hospital, Kaohsiung City, Zuoying District

IPD SHARING:
Plan to Share IPD: No